CLINICAL TRIAL: NCT02852707
Title: Physical Performance and 3D Shoulder Kinematics of Asymptomatic Unilateral/Bilateral Overhead Athletes and Non-athletes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Porto (Other)
Collaborators: University of Lisbon (Other); Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Nuno Morais, PhD student, Universidade do Porto
Other Study IDs: FADEUP_PhDPT_NunoMorais_std#1
Record Dates: First submitted 2016-07-22; First posted 2016-08-02 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Unilateral overhead throwing athletes: Volleyball attackers involved in competitive events ≥ 2 years, ≥18 years of age
  Interventions: Behavioral: Chronic exposure to unilateral overhead sports activity
- Bilateral overhead athletes: Swimmers involved in competitive events ≥ 2 years, ≥18 years of age
  Interventions: Behavioral: Chronic exposure to bilateral overhead sports activity
- Non-athletes: Persons not regularly involved in sports activities or occupational overhead tasks (e.g. construction workers), ≥18 years of age
  Interventions: Behavioral: Not exposed

INTERVENTIONS:
Behavioral: Chronic exposure to unilateral overhead sports activity — Overhead sports athletes that have been chronically exposed (≥ 2 years) predominantly to specific unilateral overhead movement patterns of the dominant extremity ("throwing arm"), such as throwing or hitting a ball ("asymmetrical overhead sports).
  Groups: Unilateral overhead throwing athletes
Behavioral: Chronic exposure to bilateral overhead sports activity — Overhead sports athletes that have been chronically exposed (≥ 2 years) predominantly to bilateral overhead movement patterns of the upper extremities, such as swimmers ("symmetrical overhead sports").
  Groups: Bilateral overhead athletes
Behavioral: Not exposed — People not engaged in regular sports competition/exercise training.
  Groups: Non-athletes

SUMMARY:
This study compares the performance and 3-dimensional shoulder kinematics between sides in unilateral overhead-throwers (volleyball attackers), bilateral overhead athletes (swimmers) and non-athletes during two physical performance measures of the upper extremity, one in an open kinetic chain position (unilateral seated shot put test) and the other in a closed kinetic chain position (upper quarter Y balance test)

DETAILED DESCRIPTION:
3-dimensional shoulder kinematics (e.g., scapular angular position/displacement) at key events of each test will be described and compared across sides and groups. For the unilateral seated shot put test, the events are based on humeral motion: a) initiation of humeral motion, b) maximal humeral flexion, c) end of humeral motion. For the upper quarter Y balance test the events are the a) initiation of free hand motion on "GO", b) maximal reach on the medial direction, c) maximal reach on superolateral direction, and d) maximal reach on the inferolateral direction (kinematics measured on the stance upper extremity). The best of 3 maximal-effort trials on each side will be used for analysis. Warm-up exercises and two submaximal practice trials will be performed for preparation for maximal efforts and familiarization with the tests. A rest period of at least one minute between trials will be given to guarantee good physiological conditions to maximally perform. Further resting time will be allowed, if necessary, upon request of the participant.

ELIGIBILITY:
Inclusion Criteria:

* Perform at least 150 degrees of arm elevation

Exclusion Criteria:

* history of shoulder dislocation
* surgery in the upper extremity ≥ 6 months
* injury in the past month
* evident abnormalities in posture and movement of the upper body quadrant
* pain at the time of testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Athletes from sports organizations involved in competitive events and non-athletes from the general community/scholarly community
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Side-to-side differences in the unilateral seated shot put test (normalized distance thrown, in centimeters) | Through study completion, an average of 1 year
  The unilateral seated shot put test consists of pushing (not throwing) at shoulder height a ~3kg medicine ball as far and forward as possible while keeping the axial skeleton in contact with a wall, knees bent at a right angle, feet flat on the floor, and the non-testing arm resting on the lap.
Side-to-side differences in the upper quarter Y balance test (normalized maximal distance reached in each direction, in centimeters) | Through study completion, an average of 1 year
  The upper quarter Y balance test is performed through the assistance of a testing device (Y-Balance Test Kit), with the subject stabilizing his/her body weight with the upper extremity being tested while performing maximal reaching efforts with the free hand in three directions: medial, superolateral, and inferolateral.

SECONDARY OUTCOMES:
Side-to-side differences in 3-dimensional scapular angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the scapula in the 3 planes of orientation: lateral/medial (upward/downward) rotation, protraction/retraction (internal/external rotation), anterior/posterior tilting.
Side-to-side differences in 3-dimensional humerus angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the humerus in the 3 planes of orientation: plane of elevation, elevation/depression, axial rotation.
Side-to-side differences in 3-dimensional thoracic angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the thorax in the 3 planes of orientation: flexion/extension, lateral rotation (inclination), axial rotation.
Side-to-side differences in the upper quarter Y balance test (total excursion, in centimeters) | Through study completion, an average of 1 year
  total excursion = sum of the 3 normalized reach distances, in centimeters
Side-to-side differences in the upper quarter Y balance test (overall performance score, in centimeters) | Through study completion, an average of 1 year
  overall performance or composite score = average score of the 3 normalized reach distances, in centimeters.

CONTACTS AND LOCATIONS:
Locations (3):
- Portugal (3):
  - Faculdade de Motricidade Humana, Universidade de Lisboa, Oeiras, Cruz-Quebrada
  - Escola Superior de Saúde, Instituto Politécnico de Leiria, Leiria
  - Faculdade de Desporto, Universidade do Porto, Porto